CLINICAL TRIAL: NCT04468191
Title: Quantifying Fatigue of the Respiratory and Swallowing Musculature in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Fatigue in Patients With Amyotrophic Lateral Sclerosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic restrictions for data collection
Sponsor: Cara Donohue (Other)
Responsible Party: Sponsor-Investigator, Cara Donohue, MA CCC-SLP/PhD Student, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20060082
Record Dates: First submitted 2020-06-22; First posted 2020-07-13 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Amyotrophic Lateral Sclerosis; Dysphagia; Dyspnea; Respiration Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Deglutition Disorders; Dyspnea; Respiration Disorders

STUDY DESIGN:
Intervention Model Description: This study will be a prospective study with randomized experimental and control conditions. Patients with ALS will undergo the experimental and control conditions in random order on two separate days within a two-week time frame.
Who Masked: Participant, Care Provider
Masking Description: During the experimental condition, expiratory muscle strength training (EMST) devices will be set to 50% of patients with ALS' highest maximum expiratory pressure from their baseline pulmonary function test assessment. During the control condition, no resistance will be added, and the loaded spring will be removed from the device. For both experimental conditions, patients with ALS will be blinded to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental, then sham (Experimental): Patients with ALS in the experimental, then sham arm will undergo an expiratory muscle strength training (EMST) session with a device set to 50% of patients with ALS' highest maximum expiratory pressure from their baseline pulmonary function test assessment during their first study visit. Then, during their second study visit, patients with ALS will undergo an EMST session with a device set to 0% resistance.
  Interventions: Device: Experimental expiratory muscle strength training (EMST); Device: Sham expiratory muscle strength training (EMST)
- Sham, then experimental (Experimental): Patients with ALS in the sham, then experimental arm will undergo an expiratory muscle strength training (EMST) session with a device set to 0% resistance during their first study visit. Then, during their second study visit, patients with ALS will undergo an EMST session with a device set to 50% of patients with ALS' highest maximum expiratory pressure from their baseline pulmonary function test assessment.
  Interventions: Device: Experimental expiratory muscle strength training (EMST); Device: Sham expiratory muscle strength training (EMST)

INTERVENTIONS:
Device: Experimental expiratory muscle strength training (EMST) — The experimental EMST will involve blowing into a device with a spring-loaded valve set to 50% of the patient with ALS' maximum expiratory pressure.
Device: Sham expiratory muscle strength training (EMST) — The sham EMST will involve blowing into a device without a spring-loaded valve (0% resistance).

SUMMARY:
Expiratory muscle strength training (EMST) is an emerging palliative intervention for prolonging pulmonary and swallow function in patients with amyotrophic lateral sclerosis (PALS), but it is unknown whether EMST may result in detrimental immediate to short-term fatigue because there is no way to measure fatigue non-invasively. This study will determine the immediate to short-term impact of EMST on objective respiratory and swallow function, whether subjective ratings of dyspnea and fatigue map to objective decompensation of respiratory and swallow function, and the ability to monitor fatigue of the respiratory and swallowing musculature non-invasively. Findings from this research study will provide preliminary evidence regarding optimal timing for PALS to complete EMST and will provide PALS and clinicians increased capabilities to monitor fatigue non-invasively.

DETAILED DESCRIPTION:
This research proposal will determine the immediate impact of expiratory muscle strength training (EMST) on fatigue of the respiratory and swallowing musculature, whether objective decompensation translates to subjective dyspnea and fatigue, and whether high resolution cervical auscultation (HRCA) signal features can noninvasively capture and characterize physiologic decompensation that relates to fatigue in patients with amyotrophic lateral sclerosis (PALS) via three Specific Aims.

Aim 1) Determine the impact of one EMST session on objective respiratory and swallow function.

Hypothesis 1) One EMST session will result in reduced pulmonary function tests (PFTs) (maximum expiratory pressure, forced vital capacity, peak cough flow) and declines in swallow function (Videofluoroscopy (VF), HRCA). PALS will have greater reductions in PFTs, and objective declines in swallow function after the experimental condition compared to the control condition.

Aim 2) Determine if objective decompensation translates to subjective ratings of dyspnea and fatigue after one EMST session.

Hypothesis 2) Subjective ratings of dyspnea and fatigue (Situational Fatigue Scale; Dyspnea ALS-15) will be associated with objective decompensation in respiratory and swallow function (PFTs, VF, HRCA) after one EMST session.

Aim 3) Investigate whether HRCA signal features analyses can non-invasively characterize immediate post-exercise physiologic changes in swallowing function that are related to fatigue.

Hypothesis 3) Pre- to post-EMST changes in HRCA signal features will be associated with physiologic changes in swallowing as measured by VF analyses.

This study will be a prospective study with randomized experimental and control conditions; and is directly related to the NIH funded research studies currently conducted in the Computational Deglutition (CD) Lab under the leadership of Dr. James Coyle and Dr. Ervin Sejdic.

Participants: 20 PALS will be recruited to undergo VF before and after undergoing the randomly ordered experimental and control conditions on two separate nonconsecutive days within a two-week time frame.

Baseline Procedures:

PALS will be instructed not to eat a meal or engage in exercise within two hours of their visit. Following consent, baseline assessment procedures be obtained. All baseline measurements of swallowing and pulmonary function will be performed before any potentially fatigue-inducing procedures are performed (i.e. exercise training).

1. The ALS functional rating scale revised (ALSFRS-R) (an instrument used to assess changes in functional status over time in PALS), will be completed.
2. Prior to completing swallowing and pulmonary measurements, PALS will complete the situational fatigue scale (SFS), which measures fatigue that results from completing functional daily activities.
3. Before undergoing swallowing and pulmonary measurements, PALS will also complete the Dyspnea ALS-15 (DALS-15), which is a measure of dyspnea that is known to be related to fatigue in PALS.
4. PALS will undergo an assessment of swallow function with concurrent recordings of videofluoroscopy (VF) and high-resolution cervical auscultation (HRCA) signals prior to undergoing PFTs to mitigate fatigue from the PFTs as a confound. VF procedures will be conducted first, because ten swallows of thin liquid are unlikely to cause fatigue of the respiratory and swallow musculature that would impact PFTs.
5. PALS will be seated upright in a chair and viewed in the lateral plane. HRCA signals will be simultaneously recorded from neck sensors (a contact microphone and accelerometer) that are attached to the anterior laryngeal framework with tape. VF and HRCA signals will be recorded onto a Labview Workstation. During each stage (pre-, post EMST) of VF, PALS will swallow ten thin liquid boluses of barium. Five liquid swallows will be a self-selected comfortable sip from a cup and five will be 3mL by spoon administered with a command to swallow. Presentation order for the liquid swallows will be randomized using a random number generator. If more than one aspiration event is observed during VF, the exam will be terminated immediately in order to ensure patient safety.
6. PFTs following VF will include maximum expiratory pressure (MEP) (measured with the MicroRPM handheld MEP device (Micro Direct Inc., Lewiston, ME)), peak cough flow (PCF) (measured with a handheld peak flow meter (BV Medical, Barrington, IL)), and FVC (measured with the Spirodoc spirometer and WinspiroPRO computer software (Medical International Research, New Berlin, WI)). All PFTs will be completed three times with PALS sitting in an upright seated position with a nose clip in line with standard PFT protocols. The highest of three measurements will be used for analyses.

EMST Training: PALS will use the EMST-150 device (Aspire Products, Gainesville, Florida) or the Philips Threshold PEP trainer (Philips Respironics, Cedar Grove, New Jersey). During the experimental condition, EMST devices will be set to 50% of PALS' highest MEP from their baseline PFT assessment. During the control condition, no resistance will be added, and the loaded spring will be removed from the device. For both experimental conditions, PALS will undergo the following standard treatment protocol:

1. PALS will complete five sets of five repetitions using an EMST device.
2. For each repetition, PALS will be instructed to take a deep breath in and blow until the valve releases.
3. Between repetitions, PALs will have 10-15 seconds of rest before the next repetition.
4. After each set, PALS will rest for one minute before completing the next set.

Post-treatment procedures: Following the EMST session with either the device set to 50% load or the sham device, PALS will undergo the same procedures (VF, HRCA, PFTs) as described above in steps 1-6 of the baseline procedures

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS defined as possible, probable, or definite by a neurologist using the El Escorial criteria
* FVC>65% predicted
* adequate cognition as defined by a score of >10 on the ALS Cognitive Behavioral Screen
* adequate labial seal for completing pulmonary function tests and expiratory muscle strength training (EMST)
* on a regular/thin liquid diet
* no allergies to barium
* not oxygen-dependent
* no tracheostomy/ mechanical ventilation
* no history of other neurological or respiratory disorders
* no history of smoking
* no history of head and neck cancer or other major head/neck surgery or radiation therapy.

Exclusion Criteria:

* FVC<65% predicted
* inadequate cognition as defined by a score of <10 on the ALS Cognitive Behavioral Screen -inadequate labial seal for completing pulmonary function tests and expiratory muscle strength training (EMST)
* not on a regular/thin liquid diet
* allergies to barium
* oxygen-dependent
* presence of tracheostomy/dependent on mechanical ventilation
* history of other neurological or respiratory disorders
* history of smoking
* history of head and neck cancer or other major head/neck surgery or radiation therapy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Change in forced vital capacity (FVC) between pre and post expiratory muscle strength training (EMST) experimental session | pre and post EMST experimental session, up to 2 weeks
  FVC is a measure of the total amount of air that can be breathed out during a pulmonary function test to measure lung function.
Change in forced vital capacity (FVC) between pre and post expiratory muscle strength training (EMST) sham session | pre and post EMST sham session, up to 2 weeks
  FVC is a measure of the total amount of air that can be breathed out during a pulmonary function test to measure lung function.
Change in peak cough flow (PCF) between pre and post expiratory muscle strength training (EMST) experimental session | pre and post EMST experimental session, up to 2 weeks
  PCF is a measure of air flow during a cough.
Change in peak cough flow (PCF) between pre and post expiratory muscle strength training (EMST) sham session | pre and post EMST sham session, up to 2 weeks
  PCF is a measure of air flow during a cough.
Change in maximum expiratory pressure (MEP) between pre and post expiratory muscle strength training (EMST) experimental session | pre and post EMST experimental session, up to 2 weeks
  Maximum expiratory pressure is a measure of strength of the respiratory muscles when breathing out
Change in maximum expiratory pressure (MEP) between pre and post expiratory muscle strength training (EMST) sham session | pre and post EMST sham session, up to 2 weeks
  Maximum expiratory pressure is a measure of strength of the respiratory muscles when breathing out
Change in temporal kinematic measures of swallowing between pre and post expiratory muscle strength training (EMST) experimental session | pre and post EMST experimental session, up to 2 weeks
  Timing measures of physiological events that occur during swallowing based on videofluoroscopic swallow studies (measured in frames per second)
Change in temporal kinematic measures of swallowing between pre and post expiratory muscle strength training (EMST) sham session | pre and post EMST sham session, up to 2 weeks
  Timing measures of physiological events that occur during swallowing based on videofluoroscopic swallow studies (measured in frames per second)
Change in spatial kinematic measures of swallowing between pre and post expiratory muscle strength training (EMST) experimental session | pre and post EMST experimental session, up to 2 weeks
  Distance measures of physiological events that occur during swallowing based on videofluoroscopic swallow studies (measured in pixels)
Change in spatial kinematic measures of swallowing between pre and post expiratory muscle strength training (EMST) sham session | pre and post EMST sham session, up to 2 weeks
  Distance measures of physiological events that occur during swallowing based on videofluoroscopic swallow studies (measured in pixels)
Change in Modified Barium Swallow Impairment Profile (MBSImP) scores of swallowing between pre and post expiratory muscle strength training (EMST) experimental session | pre and post EMST experimental session, up to 2 weeks
  The MBSImP is a standardized clinical ordinal, categorical rating tool of 17 physiological components of swallowing
Change in Modified Barium Swallow Impairment Profile (MBSImP) scores of swallowing between pre and post expiratory muscle strength training (EMST) sham session | pre and post EMST sham session, up to 2 weeks
  The MBSImP is a standardized clinical ordinal, categorical rating tool of 17 physiological components of swallowing

SECONDARY OUTCOMES:
Change in high resolution cervical auscultation (HRCA) signal features between pre and post expiratory muscle strength training (EMST) experimental session | pre and post EMST experimental session, up to 2 weeks
  Feature extraction and analyses from HRCA will be completed before and after each EMST session and compared to VF to determine whether HRCA can detect fatigue related changes in swallow function.
Change in high resolution cervical auscultation (HRCA) signal features between pre and post expiratory muscle strength training (EMST) sham session | pre and post EMST sham session, up to 2 weeks
  Feature extraction and analyses from HRCA will be completed before and after each EMST session and compared to VF to determine whether HRCA can detect fatigue related changes in swallow function.

CONTACTS AND LOCATIONS:
Overall Officials: Cara A Donohue, MA CCC-SLP, Principal Investigator — University of Pittsburgh; James L Coyle, PhD, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ball LJ, Willis A, Beukelman DR, Pattee GL. A protocol for identification of early bulbar signs in amyotrophic lateral sclerosis. J Neurol Sci. 2001 Oct 15;191(1-2):43-53. doi: 10.1016/s0022-510x(01)00623-2. PMID 11676991
- [Background] Kuhnlein P, Gdynia HJ, Sperfeld AD, Lindner-Pfleghar B, Ludolph AC, Prosiegel M, Riecker A. Diagnosis and treatment of bulbar symptoms in amyotrophic lateral sclerosis. Nat Clin Pract Neurol. 2008 Jul;4(7):366-74. doi: 10.1038/ncpneuro0853. Epub 2008 Jun 17. PMID 18560390
- [Background] da Costa Franceschini A, Mourao LF. Dysarthria and dysphagia in Amyotrophic Lateral Sclerosis with spinal onset: a study of quality of life related to swallowing. NeuroRehabilitation. 2015;36(1):127-34. doi: 10.3233/NRE-141200. PMID 25547774
- [Background] Paris G, Martinaud O, Petit A, Cuvelier A, Hannequin D, Roppeneck P, Verin E. Oropharyngeal dysphagia in amyotrophic lateral sclerosis alters quality of life. J Oral Rehabil. 2013 Mar;40(3):199-204. doi: 10.1111/joor.12019. Epub 2012 Dec 27. PMID 23278936
- [Background] Andrews JA, Meng L, Kulke SF, Rudnicki SA, Wolff AA, Bozik ME, Malik FI, Shefner JM. Association Between Decline in Slow Vital Capacity and Respiratory Insufficiency, Use of Assisted Ventilation, Tracheostomy, or Death in Patients With Amyotrophic Lateral Sclerosis. JAMA Neurol. 2018 Jan 1;75(1):58-64. doi: 10.1001/jamaneurol.2017.3339. PMID 29181534
- [Background] Plowman EK, Watts SA, Tabor L, Robison R, Gaziano J, Domer AS, Richter J, Vu T, Gooch C. Impact of expiratory strength training in amyotrophic lateral sclerosis. Muscle Nerve. 2016 Jun;54(1):48-53. doi: 10.1002/mus.24990. Epub 2016 Mar 3. PMID 26599236
- [Background] Tabor LC, Rosado KM, Robison R, Hegland K, Humbert IA, Plowman EK. Respiratory training in an individual with amyotrophic lateral sclerosis. Ann Clin Transl Neurol. 2016 Sep 1;3(10):819-823. doi: 10.1002/acn3.342. eCollection 2016 Oct. PMID 27752517
- [Background] Robison R, Tabor-Gray LC, Wymer JP, Plowman EK. Combined respiratory training in an individual with C9orf72 amyotrophic lateral sclerosis. Ann Clin Transl Neurol. 2018 Aug 21;5(9):1134-1138. doi: 10.1002/acn3.623. eCollection 2018 Sep. PMID 30250869
- [Background] Plowman EK, Tabor-Gray L, Rosado KM, Vasilopoulos T, Robison R, Chapin JL, Gaziano J, Vu T, Gooch C. Impact of expiratory strength training in amyotrophic lateral sclerosis: Results of a randomized, sham-controlled trial. Muscle Nerve. 2019 Jan;59(1):40-46. doi: 10.1002/mus.26292. Epub 2018 Nov 29. PMID 29981250
- [Background] de Almeida JP, Silvestre R, Pinto AC, de Carvalho M. Exercise and amyotrophic lateral sclerosis. Neurol Sci. 2012 Feb;33(1):9-15. doi: 10.1007/s10072-011-0921-9. Epub 2012 Jan 7. PMID 22228269
- [Background] Harkawik, R., Coyle, J.L. Exercise for better ALS management? ASHA Leader. 2012; 17(11). http://leader.pubs.asha.org/article.aspx?articleid=2292004
- [Background] Casaburi R. Principles of exercise training. Chest. 1992 May;101(5 Suppl):263S-267S. PMID 1576847
- [Background] Gibbons C, Pagnini F, Friede T, Young CA. Treatment of fatigue in amyotrophic lateral sclerosis/motor neuron disease. Cochrane Database Syst Rev. 2018 Jan 2;1(1):CD011005. doi: 10.1002/14651858.CD011005.pub2. PMID 29293261
- [Background] Dudik JM, Coyle JL, Sejdic E. Dysphagia Screening: Contributions of Cervical Auscultation Signals and Modern Signal-Processing Techniques. IEEE Trans Hum Mach Syst. 2015 Aug;45(4):465-477. doi: 10.1109/THMS.2015.2408615. PMID 26213659
- [Background] Jestrovic I, Dudik JM, Luan B, Coyle JL, Sejdic E. The effects of increased fluid viscosity on swallowing sounds in healthy adults. Biomed Eng Online. 2013 Sep 10;12:90. doi: 10.1186/1475-925X-12-90. PMID 24020398
- [Background] Dudik JM, Kurosu A, Coyle JL, Sejdic E. A statistical analysis of cervical auscultation signals from adults with unsafe airway protection. J Neuroeng Rehabil. 2016 Jan 22;13:7. doi: 10.1186/s12984-015-0110-9. PMID 26801236
- [Background] Dudik JM, Jestrovic I, Luan B, Coyle JL, Sejdic E. Characteristics of Dry Chin-Tuck Swallowing Vibrations and Sounds. IEEE Trans Biomed Eng. 2015 Oct;62(10):2456-64. doi: 10.1109/TBME.2015.2431999. Epub 2015 May 12. PMID 25974926
- [Background] Prabhu DNF, Reddy NP, Canilang EP. Neural networks for recognition of acceleration pattern during swallowing and coughing. Proceedings of 16th Annual International Conference of the IEEE Engineering in Medicine and Biology Society.1994; 1105-1106.
- [Background] Lee J, Steele CM, Chau T. Classification of healthy and abnormal swallows based on accelerometry and nasal airflow signals. Artif Intell Med. 2011 May;52(1):17-25. doi: 10.1016/j.artmed.2011.03.002. Epub 2011 May 6. PMID 21549579
- [Background] Sejdic E, Dudik JM, Kurosu A, Jestrovic I, Coyle JL. Understanding differences between healthy swallows and penetration-aspiration swallows via compressive sensing of tri-axial swallowing accelerometry signals. Proc SPIE Int Soc Opt Eng. 2014 May 23;9190:91090M. doi: 10.1117/12.2050356. PMID 25332758
- [Background] Dudik JM, Coyle JL, El-Jaroudi A, Mao ZH, Sun M, Sejdic E. Deep Learning for Classification of Normal Swallows in Adults. Neurocomputing (Amst). 2018 Apr 12;285:1-9. doi: 10.1016/j.neucom.2017.12.059. Epub 2018 Jan 31. PMID 29755210
- [Background] He Q, Perera S, Khalifa Y, Zhang Z, Mahoney AS, Sabry A, Donohue C, Coyle JL, Sejdic E. The Association of High Resolution Cervical Auscultation Signal Features With Hyoid Bone Displacement During Swallowing. IEEE Trans Neural Syst Rehabil Eng. 2019 Sep;27(9):1810-1816. doi: 10.1109/TNSRE.2019.2935302. Epub 2019 Aug 21. PMID 31443032
- [Background] Zhang Z, Perera S, Donohue C, Kurosu A, Mahoney AS, Coyle JL, Sejdic E. The Prediction of Risk of Penetration-Aspiration Via Hyoid Bone Displacement Features. Dysphagia. 2020 Feb;35(1):66-72. doi: 10.1007/s00455-019-10000-5. Epub 2019 Mar 27. PMID 30919104
- [Background] Mao S, Zhang Z, Khalifa Y, Donohue C, Coyle JL, Sejdic E. Neck sensor-supported hyoid bone movement tracking during swallowing. R Soc Open Sci. 2019 Jul 10;6(7):181982. doi: 10.1098/rsos.181982. eCollection 2019 Jul. PMID 31417694
- [Background] Donohue C, Mao S, Sejdic E, Coyle JL. Tracking Hyoid Bone Displacement During Swallowing Without Videofluoroscopy Using Machine Learning of Vibratory Signals. Dysphagia. 2021 Apr;36(2):259-269. doi: 10.1007/s00455-020-10124-z. Epub 2020 May 17. PMID 32419103
- [Background] Khalifa Y, Donohue C, Coyle JL, Sejdic E. Upper Esophageal Sphincter Opening Segmentation With Convolutional Recurrent Neural Networks in High Resolution Cervical Auscultation. IEEE J Biomed Health Inform. 2021 Feb;25(2):493-503. doi: 10.1109/JBHI.2020.3000057. Epub 2021 Feb 5. PMID 32750928
- [Background] Sabry A, Shitong M, Mahoney A, Khalifa Y, Sejdic E, Coyle J. Automatic estimation of laryngeal vestibular closure duration using high resolution cervical auscultation signals. Presentation at the American Speech-Language Hearing Association Convention, Orlando, FL. 2019.
- [Background] Donohue C, Zhenwei Z, Mahoney A, Perera S, Sejdic E, Coyle J. Do machine ratings of hyoid bone displacement during videofluoroscopy match clinician ratings using the MBSImP? Presentation at the American Speech-Language Hearing Association Annual Meeting, Boston, MA. November 2018.
- [Background] Sabry A, Mahoney A, Perera S, Sejdic E, Coyle J. Are HRCA signal features associated with clinical ratings of pharyngeal residue using the MBSImP? Presentation at the Dysphagia Research Society Annual Meeting, San Diego, CA. March 2019.
- [Background] Donohue C, Khalifa Y, Perera S, Sejdic E, Coyle JL. How Closely do Machine Ratings of Duration of UES Opening During Videofluoroscopy Approximate Clinician Ratings Using Temporal Kinematic Analyses and the MBSImP? Dysphagia. 2021 Aug;36(4):707-718. doi: 10.1007/s00455-020-10191-2. Epub 2020 Sep 21. PMID 32955619
- [Background] Kurosu A, Coyle JL, Dudik JM, Sejdic E. Detection of Swallow Kinematic Events From Acoustic High-Resolution Cervical Auscultation Signals in Patients With Stroke. Arch Phys Med Rehabil. 2019 Mar;100(3):501-508. doi: 10.1016/j.apmr.2018.05.038. Epub 2018 Jul 30. PMID 30071198
- [Background] Donohue C, Khalifa Y, Perera S, Sejdic E, Coyle JL. A Preliminary Investigation of Whether HRCA Signals Can Differentiate Between Swallows from Healthy People and Swallows from People with Neurodegenerative Diseases. Dysphagia. 2021 Aug;36(4):635-643. doi: 10.1007/s00455-020-10177-0. Epub 2020 Sep 5. PMID 32889627
- [Background] Hiramatsu T, Kataoka H, Osaki M, Hagino H. Effect of aging on oral and swallowing function after meal consumption. Clin Interv Aging. 2015 Jan 9;10:229-35. doi: 10.2147/CIA.S75211. eCollection 2015. PMID 25624755
- [Background] Kays SA, Hind JA, Gangnon RE, Robbins J. Effects of dining on tongue endurance and swallowing-related outcomes. J Speech Lang Hear Res. 2010 Aug;53(4):898-907. doi: 10.1044/1092-4388(2009/09-0048). PMID 20689047
- [Background] Kim DG, Hong YH, Shin JY, Lee KW, Park KS, Seong SY, Sung JJ. Pattern of Respiratory Deterioration in Sporadic Amyotrophic Lateral Sclerosis According to Onset Lesion by Using Respiratory Function Tests. Exp Neurobiol. 2015 Dec;24(4):351-7. doi: 10.5607/en.2015.24.4.351. Epub 2015 Nov 4. PMID 26713082
- [Background] Schmidt EP, Drachman DB, Wiener CM, Clawson L, Kimball R, Lechtzin N. Pulmonary predictors of survival in amyotrophic lateral sclerosis: use in clinical trial design. Muscle Nerve. 2006 Jan;33(1):127-32. doi: 10.1002/mus.20450. PMID 16258948
- [Background] Suarez AA, Pessolano FA, Monteiro SG, Ferreyra G, Capria ME, Mesa L, Dubrovsky A, De Vito EL. Peak flow and peak cough flow in the evaluation of expiratory muscle weakness and bulbar impairment in patients with neuromuscular disease. Am J Phys Med Rehabil. 2002 Jul;81(7):506-11. doi: 10.1097/00002060-200207000-00007. PMID 12131177
- [Background] Baumann F, Henderson RD, Morrison SC, Brown M, Hutchinson N, Douglas JA, Robinson PJ, McCombe PA. Use of respiratory function tests to predict survival in amyotrophic lateral sclerosis. Amyotroph Lateral Scler. 2010;11(1-2):194-202. doi: 10.3109/17482960902991773. PMID 19452343
- [Background] Vogt S, Petri S, Dengler R, Heinze HJ, Vielhaber S. Dyspnea in Amyotrophic Lateral Sclerosis: Rasch-Based Development and Validation of a Patient-Reported Outcome (DALS-15). J Pain Symptom Manage. 2018 Nov;56(5):736-745.e2. doi: 10.1016/j.jpainsymman.2018.08.009. Epub 2018 Aug 24. PMID 30145215
- [Background] Homepage - ALS Association. ALSA.org. http://www.alsa.org/. Accessed April 10, 2019.
- [Background] Wilkins T, Gillies RA, Thomas AM, Wagner PJ. The prevalence of dysphagia in primary care patients: a HamesNet Research Network study. J Am Board Fam Med. 2007 Mar-Apr;20(2):144-50. doi: 10.3122/jabfm.2007.02.060045. PMID 17341750
- [Background] Barer DH. The natural history and functional consequences of dysphagia after hemispheric stroke. J Neurol Neurosurg Psychiatry. 1989 Feb;52(2):236-41. doi: 10.1136/jnnp.52.2.236. PMID 2564884
- [Background] Flowers HL, Silver FL, Fang J, Rochon E, Martino R. The incidence, co-occurrence, and predictors of dysphagia, dysarthria, and aphasia after first-ever acute ischemic stroke. J Commun Disord. 2013 May-Jun;46(3):238-48. doi: 10.1016/j.jcomdis.2013.04.001. Epub 2013 Apr 12. PMID 23642855
- [Background] Gordon C, Hewer RL, Wade DT. Dysphagia in acute stroke. Br Med J (Clin Res Ed). 1987 Aug 15;295(6595):411-4. doi: 10.1136/bmj.295.6595.411. PMID 3115478
- [Background] Alagiakrishnan K, Bhanji RA, Kurian M. Evaluation and management of oropharyngeal dysphagia in different types of dementia: a systematic review. Arch Gerontol Geriatr. 2013 Jan-Feb;56(1):1-9. doi: 10.1016/j.archger.2012.04.011. Epub 2012 May 19. PMID 22608838
- [Background] Garcia-Peris P, Paron L, Velasco C, de la Cuerda C, Camblor M, Breton I, Herencia H, Verdaguer J, Navarro C, Clave P. Long-term prevalence of oropharyngeal dysphagia in head and neck cancer patients: Impact on quality of life. Clin Nutr. 2007 Dec;26(6):710-7. doi: 10.1016/j.clnu.2007.08.006. Epub 2007 Oct 22. PMID 17954003
- [Background] Skoretz SA, Flowers HL, Martino R. The incidence of dysphagia following endotracheal intubation: a systematic review. Chest. 2010 Mar;137(3):665-73. doi: 10.1378/chest.09-1823. PMID 20202948
- [Background] Martin-Harris B. Clinical implications of respiratory-swallowing interactions. Curr Opin Otolaryngol Head Neck Surg. 2008 Jun;16(3):194-9. doi: 10.1097/MOO.0b013e3282febd4b. PMID 18475070
- [Background] Larkindale J, Yang W, Hogan PF, Simon CJ, Zhang Y, Jain A, Habeeb-Louks EM, Kennedy A, Cwik VA. Cost of illness for neuromuscular diseases in the United States. Muscle Nerve. 2014 Mar;49(3):431-8. doi: 10.1002/mus.23942. Epub 2014 Jan 28. PMID 23836444
- [Background] Lechtzin N, Wiener CM, Clawson L, Chaudhry V, Diette GB. Hospitalization in amyotrophic lateral sclerosis: causes, costs, and outcomes. Neurology. 2001 Mar 27;56(6):753-7. doi: 10.1212/wnl.56.6.753. PMID 11274310
- [Background] Enoka RM, Duchateau J. Muscle fatigue: what, why and how it influences muscle function. J Physiol. 2008 Jan 1;586(1):11-23. doi: 10.1113/jphysiol.2007.139477. Epub 2007 Aug 16. PMID 17702815
- [Background] Hunter SK, Duchateau J, Enoka RM. Muscle fatigue and the mechanisms of task failure. Exerc Sport Sci Rev. 2004 Apr;32(2):44-9. doi: 10.1097/00003677-200404000-00002. PMID 15064647
- [Background] Kirkinezos IG, Hernandez D, Bradley WG, Moraes CT. Regular exercise is beneficial to a mouse model of amyotrophic lateral sclerosis. Ann Neurol. 2003 Jun;53(6):804-7. doi: 10.1002/ana.10597. PMID 12783429
- [Background] Mahoney DJ, Rodriguez C, Devries M, Yasuda N, Tarnopolsky MA. Effects of high-intensity endurance exercise training in the G93A mouse model of amyotrophic lateral sclerosis. Muscle Nerve. 2004 May;29(5):656-62. doi: 10.1002/mus.20004. PMID 15116368
- [Background] Aitkens SG, McCrory MA, Kilmer DD, Bernauer EM. Moderate resistance exercise program: its effect in slowly progressive neuromuscular disease. Arch Phys Med Rehabil. 1993 Jul;74(7):711-5. doi: 10.1016/0003-9993(93)90031-5. PMID 8328892
- [Background] Dal Bello-Haas V, Florence JM. Therapeutic exercise for people with amyotrophic lateral sclerosis or motor neuron disease. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD005229. doi: 10.1002/14651858.CD005229.pub3. PMID 23728653
- [Background] Kent-Braun JA, Miller RG. Central fatigue during isometric exercise in amyotrophic lateral sclerosis. Muscle Nerve. 2000 Jun;23(6):909-14. doi: 10.1002/(sici)1097-4598(200006)23:63.0.co;2-v. PMID 10842267
- [Background] Vucic S, Cheah BC, Kiernan MC. Maladaptation of cortical circuits underlies fatigue and weakness in ALS. Amyotroph Lateral Scler. 2011 Nov;12(6):414-20. doi: 10.3109/17482968.2011.597403. Epub 2011 Aug 11. PMID 21830989
- [Background] Kent-Braun JA, Fitts RH, Christie A. Skeletal muscle fatigue. Compr Physiol. 2012 Apr;2(2):997-1044. doi: 10.1002/cphy.c110029. PMID 23798294
- [Background] Tabor L, Gaziano J, Watts S, Robison R, Plowman EK. Defining Swallowing-Related Quality of Life Profiles in Individuals with Amyotrophic Lateral Sclerosis. Dysphagia. 2016 Jun;31(3):376-82. doi: 10.1007/s00455-015-9686-2. Epub 2016 Feb 2. PMID 26837611
- [Background] Luchesi KF, Campos BM, Mituuti CT. Identification of swallowing disorders: the perception of patients with neurodegenerative diseases. Codas. 2018 Nov 29;30(6):e20180027. doi: 10.1590/2317-1782/20182018027. English, Portuguese. PMID 30517269
- [Background] Roth EJ, Stenson KW, Powley S, Oken J, Primack S, Nussbaum SB, Berkowitz M. Expiratory muscle training in spinal cord injury: a randomized controlled trial. Arch Phys Med Rehabil. 2010 Jun;91(6):857-61. doi: 10.1016/j.apmr.2010.02.012. PMID 20510974
- [Background] Troche MS, Okun MS, Rosenbek JC, Musson N, Fernandez HH, Rodriguez R, Romrell J, Pitts T, Wheeler-Hegland KM, Sapienza CM. Aspiration and swallowing in Parkinson disease and rehabilitation with EMST: a randomized trial. Neurology. 2010 Nov 23;75(21):1912-9. doi: 10.1212/WNL.0b013e3181fef115. PMID 21098406
- [Background] Neves LF, Reis MH, Plentz RD, Matte DL, Coronel CC, Sbruzzi G. Expiratory and expiratory plus inspiratory muscle training improves respiratory muscle strength in subjects with COPD: systematic review. Respir Care. 2014 Sep;59(9):1381-8. doi: 10.4187/respcare.02793. Epub 2014 Apr 29. PMID 24782553
- [Background] Patchett KK, Hausenblas HA, Christine M. Expiratory Muscle Strength Training for Dysphagia in Chronic Obstructive Pulmonary Disease: A Meta-analysis and Systematic Review. 2017;(August 2015).
- [Background] Ferreira GD, Costa AC, Plentz RD, Coronel CC, Sbruzzi G. Respiratory training improved ventilatory function and respiratory muscle strength in patients with multiple sclerosis and lateral amyotrophic sclerosis: systematic review and meta-analysis. Physiotherapy. 2016 Sep;102(3):221-8. doi: 10.1016/j.physio.2016.01.002. Epub 2016 Mar 26. PMID 27026167
- [Background] Park JS, Oh DH, Chang MY, Kim KM. Effects of expiratory muscle strength training on oropharyngeal dysphagia in subacute stroke patients: a randomised controlled trial. J Oral Rehabil. 2016 May;43(5):364-72. doi: 10.1111/joor.12382. Epub 2016 Jan 24. PMID 26803525
- [Background] Hegland KW, Davenport PW, Brandimore AE, Singletary FF, Troche MS. Rehabilitation of Swallowing and Cough Functions Following Stroke: An Expiratory Muscle Strength Training Trial. Arch Phys Med Rehabil. 2016 Aug;97(8):1345-51. doi: 10.1016/j.apmr.2016.03.027. Epub 2016 Apr 26. PMID 27130637
- [Background] Hutcheson KA, Barrow MP, Plowman EK, Lai SY, Fuller CD, Barringer DA, Eapen G, Wang Y, Hubbard R, Jimenez SK, Little LG, Lewin JS. Expiratory muscle strength training for radiation-associated aspiration after head and neck cancer: A case series. Laryngoscope. 2018 May;128(5):1044-1051. doi: 10.1002/lary.26845. Epub 2017 Aug 22. PMID 28833185
- [Background] Pinto S, Swash M, de Carvalho M. Respiratory exercise in amyotrophic lateral sclerosis. Amyotroph Lateral Scler. 2012 Jan;13(1):33-43. doi: 10.3109/17482968.2011.626052. PMID 22214352
- [Background] Malatra I. Respiratory Muscle Fatigue and the Effects on Swallowing. ProQuest. 2016.
- [Background] Steele CM, Cichero JA. Physiological factors related to aspiration risk: a systematic review. Dysphagia. 2014 Jun;29(3):295-304. doi: 10.1007/s00455-014-9516-y. Epub 2014 Feb 23. PMID 24562507
- [Background] Donohue C, Coyle JL. Impact of respiratory interventions on pulmonary, cough, and swallowing in ALS. ASHA Perspectives. Under review.
- [Background] Carvalho DV, Santos RMS, Magalhaes HC, Souza MS, Christo PP, Almeida-Leite CM, Scalzo PL. Can fatigue predict walking capacity of patients with Parkinson's disease? Arq Neuropsiquiatr. 2020 Feb;78(2):70-75. doi: 10.1590/0004-282X20190136. PMID 32159720
- [Background] Manty M, de Leon CF, Rantanen T, Era P, Pedersen AN, Ekmann A, Schroll M, Avlund K. Mobility-related fatigue, walking speed, and muscle strength in older people. J Gerontol A Biol Sci Med Sci. 2012 May;67(5):523-9. doi: 10.1093/gerona/glr183. Epub 2011 Oct 19. PMID 22016363
- [Background] Dalgas U, Langeskov-Christensen M, Skjerbaek A, Jensen E, Baert I, Romberg A, Santoyo Medina C, Gebara B, Maertens de Noordhout B, Knuts K, Bethoux F, Rasova K, Severijns D, Bibby BM, Kalron A, Norman B, Van Geel F, Wens I, Feys P. Is the impact of fatigue related to walking capacity and perceived ability in persons with multiple sclerosis? A multicenter study. J Neurol Sci. 2018 Apr 15;387:179-186. doi: 10.1016/j.jns.2018.02.026. Epub 2018 Feb 16. PMID 29571860
- [Background] Vogt S, Schreiber S, Pfau G, Kollewe K, Heinze HJ, Dengler R, Petri S, Vielhaber S, Brinkers M. Dyspnea as a Fatigue-Promoting Factor in ALS and the Role of Objective Indicators of Respiratory Impairment. J Pain Symptom Manage. 2020 Aug;60(2):430-438.e1. doi: 10.1016/j.jpainsymman.2020.02.021. Epub 2020 Mar 5. PMID 32145336
- [Background] Yang CM, Wu CH. The situational fatigue scale: a different approach to measuring fatigue. Qual Life Res. 2005 Jun;14(5):1357-62. doi: 10.1007/s11136-004-5680-0. PMID 16047510
- [Background] Moore VC. Spirometry: Step by step. Breathe, 2012; 8(3), 233-240. https://doi.org/10.1183/20734735.0021711
- [Background] Cheung HJ, Cheung L. Coaching patients during pulmonary function testing: A practical guide. Can J Respir Ther. 2015 Summer;51(3):65-8. PMID 26283871
- [Background] Duncan P, Richards L, Wallace D, Stoker-Yates J, Pohl P, Luchies C, Ogle A, Studenski S. A randomized, controlled pilot study of a home-based exercise program for individuals with mild and moderate stroke. Stroke. 1998 Oct;29(10):2055-60. doi: 10.1161/01.str.29.10.2055. PMID 9756581
- [Background] VanSwearingen JM, Perera S, Brach JS, Cham R, Rosano C, Studenski SA. A randomized trial of two forms of therapeutic activity to improve walking: effect on the energy cost of walking. J Gerontol A Biol Sci Med Sci. 2009 Nov;64(11):1190-8. doi: 10.1093/gerona/glp098. Epub 2009 Jul 30. PMID 19643842
- [Background] Brach JS, Van Swearingen JM, Perera S, Wert DM, Studenski S. Motor learning versus standard walking exercise in older adults with subclinical gait dysfunction: a randomized clinical trial. J Am Geriatr Soc. 2013 Nov;61(11):1879-86. doi: 10.1111/jgs.12506. Epub 2013 Oct 28. PMID 24219189
- [Background] Weiner DK, Gentili A, Rossi M, Coffey-Vega K, Rodriguez KL, Hruska KL, Hausmann L, Perera S. Aging Back Clinics-a Geriatric Syndrome Approach to Treating Chronic Low Back Pain in Older Adults: Results of a Preliminary Randomized Controlled Trial. Pain Med. 2020 Feb 1;21(2):274-290. doi: 10.1093/pm/pnz179. PMID 31503275
- [Background] Resnick J, Gupta N, Wagner J, Costa G, Cruz RJ Jr, Martin L, Koritsky DA, Perera S, Matarese L, Eid K, Schuster B, Roberts M, Greenspan S, Abu-Elmagd K. Skeletal integrity and visceral transplantation. Am J Transplant. 2010 Oct;10(10):2331-40. doi: 10.1111/j.1600-6143.2010.03245.x. Epub 2010 Sep 3. PMID 20825384